CLINICAL TRIAL: NCT05673018
Title: REACH Study: Galleri® in the Medicare Population.
Brief Title: Galleri® in the Medicare Population.
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: GRAIL, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: GRAIL-MA-002
Record Dates: First submitted 2022-12-07; First posted 2023-01-05 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-02

CONDITIONS: Cancer
Keywords: ctDNA, Circulating tumor DNA, Screening, Cancer
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Intervention Model Description: The parallel arm is a passively-enrolled contemporaneous comparator cohort of Medicare beneficiaries who receive usual care without MCED screening.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (2):
- (Galleri + UC) (Experimental): Medicare beneficiaries who receive the Galleri test plus usual care (Galleri + UC).
  Interventions: Device: Multi-Cancer Early Detection Test (Galleri®)
- (UC) alone (No Intervention): Passively-enrolled Contemporaneous Comparator Arm of Medicare beneficiaries who receive usual care (UC) alone.

INTERVENTIONS:
Device: Multi-Cancer Early Detection Test (Galleri®) — Blood collection and multi-cancer early detection testing with return of results.
  Arms: (Galleri + UC)

SUMMARY:
This multi-center comparative prospective cohort study is designed to assess the real world clinical impact, including safety and test performance, of Galleri®, a blood-based multi-cancer early detection (MCED) test. The study will seek enrollment that is representative of the Medicare population.

ELIGIBILITY:
Inclusion Criteria:

For Galleri + UC (Galleri-Tested Arm):

Participants are eligible to be included in the study only if all of the following criteria apply:

* Aged ≥50 years with Medicare coverage, including Traditional Medicare (Part A & B or Dual Eligibles) or Medicare Advantage.
* Capable of giving informed consent that is legally effective (consent provided by a legally authorized representative is not permitted in this protocol).

For UC (Not Galleri-tested Arm):

Participants are eligible to be included in the study only if all of the following criteria apply:

* Aged ≥ 50 years with Medicare coverage, including Traditional Medicare (Part A & B or Dual Eligibles) or Medicare Advantage.
* Have had ≥ 1 UC visit

Exclusion Criteria:

For Galleri + UC (Galleri-Tested Arm):

* Evidence of having had a previous MCED test (including but not limited to the Galleri test, e.g. CancerSeek, PanSeer). Participation in a study such as GRAIL's STRIVE study where results were not returned is not an exclusion criterion.
* Undergoing clinical evaluation for suspicion of cancer within 6 months prior to enrollment. Personal history of hematologic malignancy and/or invasive solid tumor (excluding non-metastatic basal cell carcinoma and squamous cell carcinoma of the skin):

  1. Diagnosed ≤3 years before expected enrollment date and/or
  2. Diagnosed >3 years before expected enrollment date and never treated and/or
  3. Currently undergoing active cancer management (not including adjuvant hormone therapy for breast or prostate cancer).
* Current pregnancy.
* Individuals who are currently inpatients at a participating site.
* Individuals who are not willing or able to comply with the protocol procedures.
* Individuals who are not currently registered patients at a participating center.
* Previous or current employees or contractors of GRAIL.

For UC (Not Galleri-tested Arm):

* Evidence of having had a previous MCED test (including but not limited to the Galleri test, eg.CancerSeek, PanSeer). Participation in a study such as GRAIL's STRIVE study where results were not returned is not an exclusion criterion.
* Undergoing clinical evaluation for suspicion of cancer.
* Personal history of hematologic malignancy and/or invasive solid tumor (not including non-metastatic basal cell carcinoma and squamous cell carcinoma of the skin):

  1. Diagnosed ≤3 years before expected enrollment date and/or
  2. Diagnosed >3 years before expected enrollment date and never treated and/or
  3. Currently undergoing active cancer management (not including adjuvant hormone therapy for breast or prostate cancer).
* Current pregnancy.
* Individuals who are currently inpatients at a participating site.

Min Age: 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50000 (Estimated)
Dates: Start 2024-07-12 (Actual); Primary Completion 2030-09 (Estimated); Study Completion 2030-09 (Estimated)

PRIMARY OUTCOMES:
Incidence rates of stage IV cancers | Up to 3 Years

SECONDARY OUTCOMES:
Safety: Number and type of invasive procedures performed to evaluate a cancer signal detected test result | Up to 3 Years
Galleri test performance in the Galleri + UC arm | Up to 3 Years
Adherence to guideline-recommended cancer screening in the Galleri+UC arm and UC arm over time | Up to 3 Years
Healthcare resource utilization associated with cancer diagnostic evaluations in the Galleri+UC arm and UC arm | Up to 3 Years

CONTACTS AND LOCATIONS:
Locations (47):
- United States (47):
  - Sutter Valley Hospitals Auburn, Auburn, California
  - Sutter Valley Hospitals Davis, Davis, California
  - Sutter Valley Hospitals Elk Grove, Elk Grove, California
  - Long Beach Memorial Orange Coast, Fountain Valley, California
  - Long Beach Memorial Saddleback, Laguna Hills, California
  - Long Beach Memorial Atlantic, Long Beach, California
  - Sutter Valley Hospitals Modesto, Modesto, California
  - Sutter Valley Hospitals PAMF Sutter, Palo Alto, California
  - Sutter Valley Hospitals Roseville, Roseville, California
  - Sutter Valley Hospitals Alhambra, Sacramento, California
  - Sutter Valley Hospitals Capitol Pavilion, Sacramento, California
  - University of California San Francisco Health System, San Francisco, California
  - Sutter Valley Hospitals Santa Barbara, Santa Barbara, California
  - Sutter Valley Hospitals PAMF Santa Cruz, Santa Cruz, California
  - Sutter Health Santa Rosa, Santa Rosa, California
  - Sutter Valley Hospitals PAMF Sunnyvale, Sunnyvale, California
  - Sutter Valley Hospitals Fairfield, Vallejo, California
  - Morehouse School of Medicine Atlanta, Atlanta, Georgia
  - Morehouse School of Medicine Lee Street, Atlanta, Georgia
  - Morehouse School of Medicine Princeton Lakes, Atlanta, Georgia
  - Morehouse School of Medicine East Point, Atlanta, Georgia
  - Community Health Network Anderson, Anderson, Indiana
  - Community Health Network North, Fishers, Indiana
  - Community Health Network East, Indianapolis, Indiana
  - Community Health Network South, Indianapolis, Indiana
  - Community Health Network Kokomo, Kokomo, Indiana
  - Ochsner Health Bocage, Baton Rouge, Louisiana
  - Ochsner Health Grove, Baton Rouge, Louisiana
  - Ochsner Health Covington, Covington, Louisiana
  - Ochsner Health St. Tammany Parish, Covington, Louisiana
  - Ochsner Health STCC, Covington, Louisiana
  - Ochsner Health Kenner, Kenner, Louisiana
  - Ochsner Health Lafayette, Lafayette, Louisiana
  - Ochsner Health Westbank, Marrero, Louisiana
  - Ochsner Health Lafreniere, Metairie, Louisiana
  - Ochsner Health Benson, New Orleans, Louisiana
  - Mercy Health - Springfield, Springfield, Missouri
  - Mercy Health St. Louis, St Louis, Missouri
  - OHSU CEDAR Clinical Trials Beaverton, Beaverton, Oregon
  - OHSU CEDAR Clinical Trials Orenco, Hillsboro, Oregon
  - OHSU CEDAR Clinical Trials Portland, Portland, Oregon
  - OHSU CEDAR Clinical Trials Richmond, Portland, Oregon
  - Geisinger Bloomsburg Hospital, Bloomsburg, Pennsylvania
  - HCA Healthcare Brentwood, Brentwood, Tennessee
  - HCA Healthcare Centennial, Nashville, Tennessee
  - HCA Healthcare Nashville, Nashville, Tennessee
  - West Virginia University Health System, Morgantown, West Virginia